CLINICAL TRIAL: NCT01575496
Title: Transcranial Direct Current Stimulation (tDCS) for the Treatment of Chronic Subjective Tinnitus
Brief Title: Transcranial Direct Current Stimulation (tDCS) for the Treatment of Tinnitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, David Benninger, MD, Principal Investigator, Head of Neurophysiology Laboratory, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIV-12-02-004761
Record Dates: First submitted 2012-04-10; First posted 2012-04-11 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Tinnitus
Keywords: Tinnitus; Transcranial direct current stimulation; Transcranial magnetic stimulation
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Active tDCS (Active Comparator): Subjects will receive 20 minutes of active tDCS.
  Interventions: Device: BrainSTIM Transcranial Stimulator
- Sham tDCS (Sham Comparator): Subjects will receive 20 minutes of sham tDCS.
  Interventions: Device: BrainSTIM Transcranial Stimulator

INTERVENTIONS:
Device: BrainSTIM Transcranial Stimulator — Cathodal stimulation of the auditory cortex with an anode (reference electrode) over the prefrontal cortex. Stimulation will be applied for 20 minutes at 2 mA.
  Other Names: Cathodal tDCS; Bilateral tDCS; Direct current stimulator; Transcranial stimulator
  Arms: Active tDCS
Device: BrainSTIM Transcranial Stimulator — Sham tDCS sessions will last 20 minutes.
  Other Names: Sham stimulation; Direct current stimulator; Transcranial stimulator
  Arms: Sham tDCS

SUMMARY:
The purpose of this study is to determine if repeated sessions of transcranial direct current stimulation (tDCS) are effective for treating chronic subjective tinnitus. Previous studies have reported brief improvements in tinnitus after safe and noninvasive stimulation of the auditory cortex or limbic system. The investigators hypothesize that a greater improvement in tinnitus will be achieved following repeated sessions of tDCS that target both auditory and limbic systems.

DETAILED DESCRIPTION:
Subjective tinnitus is a distressing condition characterized by the sensation of sound or noise in the absence of internal or external stimuli. Research indicates that tinnitus may develop due to maladaptive plastic changes in the auditory cortex and limbic system. These changes can be targeted using safe and noninvasive brain stimulation techniques like transcranial direct current stimulation (tDCS). TDCS alters the excitability of the cortex using a weak direct current and may lead to long-term plastic changes, making it a potential therapeutic tool for the treatment of tinnitus.

Transient improvements in tinnitus have been reported after inhibitory stimulation of the auditory cortex and after excitatory stimulation of the prefrontal cortex, however the effects of a combined stimulation paradigm remain unknown. The investigators hypothesize that a cumulative effect will be observed following repeated sessions of tDCS by modulating both the excitability of the auditory cortex and prefrontal cortex.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years
* Chronic tinnitus for at least 1 year
* Diagnosis of chronic subjective non-pulsatile tinnitus
* Age-adjusted normal (sensorineural) hearing
* Score of 25 or above on the Mini-mental state examination (MMSE)
* Must comply with use of contraceptives during interventions

Exclusion Criteria:

* Objective tinnitus
* Concurrent treatment for tinnitus
* Prior exposure to transcranial direct current stimulation (tDCS)
* Electronic implants or metallic objects in body, including cardiac pacemakers, cochlear implants, implanted medical pump, metal plate in skull, metal implant in the skull or eyes (other than dental appliances or fillings)
* Skin conditions where electrodes will be applied
* Major neurological co-morbidities
* History of epilepsy and/or seizures
* Pregnancy and/or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI; Newman, Jacobson, & Spitzer, 1996; French version: Ghulyan-Bédikian et al., 2010) | Baseline, 1 month after last intervention
  Assesses the change in tinnitus from baseline to 1 month after intervention.

SECONDARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | Baseline, session 5 (day 5), 1 and 3 months after the last intervention
  Assesses change in tinnitus from baseline to follow-up periods post interventions.
Visual Analogue Scales (VAS) of perceived tinnitus loudness and distress | Baseline, before and after each intervention, 1 and 3 months after the last intervention
  Self assessment of tinnitus loudness and tinnitus distress.
Hospital Anxiety and Depression Scale (HAD) | Baseline, 1 month after intervention
  Assesses anxiety and depression.
Subjective Tinnitus Severity Scale (STSS) | Baseline, session 5 (day 5), 1 and 3 months after the last intervention
  Assesses tinnitus severity.
Clinical Global Impression Scale (CGI) | Session 5 (day 5), 1 and 3 months after the last intervention
  Patient rating of worsening/improvement in condition following interventions.

CONTACTS AND LOCATIONS:
Overall Officials: David Benninger, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Department of Neurology, Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland